CLINICAL TRIAL: NCT02997787
Title: Neutrophil to Lymphocyte Ratio and Platelet to Lymphocyte Ratio Can Be Useful Markers for Distinguishing Uterine Adenomyosis and Leiomyoma
Brief Title: New Inflammation Markers for Distinguishing Uterine Adenomyosis and Leiomyoma
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf MADENDAG, Director, Kayseri Education and Research Hospital
Other Study IDs: 2016/525
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Adenomyosis; Leiomyoma; Inflammation
Keywords: adenomyosis; leiomyoma; neutrophil to lymphocyte ratio; platelet to lymphocyte ratio
MeSH Terms: conditions — Adenomyosis; Leiomyoma; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- adenomyosis: First group called adenomyosis was consisted of patients who were pathologically diagnosed pure adenomyosis after hysterectomy
- leiomyoma: Second group called leiomyoma was consisted of patients who were pathologically diagnosed pure leiomyoma after hysterectomy
- control: Third group called control group was consisted of healthy patients who were pathologically diagnosed no neoplasm after hysterectomy

SUMMARY:
Both pelvic masses and preoperative diagnosis of them have still continued as an important investigation subject. It is important to discriminate the diagnoses of leiomyoma and adenomyosis before operation especially among infertile patients. Neoplasms can alter systemic or local immune response in their originating area.Neutrophil to lymphocyte ratio (NLR) and platelet to lymphocyte ratio (PLR) can be readily determined by using of complete blood counter test (CBC). A high NLR has been shown in systemic inflammation, some gynecologic and gastrointestinal cancers and some cardiovascular diseases.

The investigators aim to investigate using new inflammation markers, NLR and PLR, whether they are useful to discriminate between adenomyosis and leiomyoma. As far as is known, there have been no previous reports about the association among NLR, PLR, adenomyosis and leiomyoma.

DETAILED DESCRIPTION:
A retrospective cross-sectional study was conducted at the Kayseri Education and Research Hospital, Department of Obstetrics and Gynecology, Kayseri, Turkey, between January 2016 and October 2016.

Approval of the Institutional Review Board of Kayseri Erciyes University the Faculty of Medicine was obtained in advance (2016/525).

Exclusion criteria were as fallows; diabetes mellitus, metabolic disorder, acute or chronic infection disease, hypertension, acute coroner artery disease, connective tissue disorder, vasculitis, inflammatory bowel disease, tobacco and alcohol use, renal failure, hepatitis, patients using corticosteroid drug and patients underwent blood transfusion within three months. The investigators reviewed a database of 386 patients who were referred for abnormal uterine bleeding resistant to medical treatment or detected pelvic mass in postmenopausal and premenopausal period and underwent hysterectomy in our department. The investigators are capable of including 196 patients in the present study because of exclusion criteria.

There were three groups in our study. First group called adenomyosis was consisted of patients who were pathologically diagnosed pure adenomyosis after hysterectomy. Second group called leiomyoma was consisted of patients who were pathologically diagnosed pure leiomyoma after hysterectomy. Third group called control group was consisted of healthy patients who were pathologically diagnosed no neoplasm after hysterectomy.

In order to evaluate serum levels of hemoglobin, leukocytes, neutrophil, lymphocyte, platelet and CA125, the investigators obtained data analysis measured preoperatively from venous blood samples of all subjects. The NLR was defined as the absolute neutrophil count divided by the absolute lymphocyte count and the PLR was defined as the absolute platelet count divided by the absolute lymphocyte count.

ELIGIBILITY:
Inclusion Criteria:

* 386 patients who were referred for abnormal uterine bleeding resistant to medical treatment or detected pelvic mass in postmenopausal and premenopausal period and underwent hysterectomy in our department were evaluated. However 196 of those patients were included in the present study because of exclusion criteria.

Exclusion Criteria:

* Exclusion criteria were as fallows; diabetes mellitus, metabolic disorder, acute or chronic infection disease, hypertension, acute coroner artery disease, connective tissue disorder, vasculitis, inflammatory bowel disease, tobacco and alcohol use, renal failure, hepatitis, patients using corticosteroid drug and patients underwent blood transfusion within three months.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There were three groups in our study. First group called adenomyosis was consisted of patients who were pathologically diagnosed pure adenomyosis after hysterectomy. Second group called leiomyoma was consisted of patients who were pathologically diagnosed pure leiomyoma after hysterectomy. Third group called control group was consisted of healthy patients who were pathologically diagnosed no neoplasm after hysterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measured serum inflammatory markers among groups by complete blood count | 3 months
  Those markers are neutrophil, lymphocyte and platelet count.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Madendag, Principal Investigator — Kayseri Education and Research Hospital